CLINICAL TRIAL: NCT01360073
Title: Association Between Low Dose Acetylsalicylic Acid (ASA) and Proton Pump Inhibitors and Risk of Acute Myocardial Infarction or Coronary Heart Disease Death - Nested Case Control Analyses in a Cohort of Patients With Acute Serious Coronary Heart Disease
Brief Title: Association Between Low Dose Acetylsalicylic Acid (ASA) and Proton Pump Inhibitors and Risk of Acute Myocardial Infarction or Coronary Heart Disease Death
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D961FN00007
Record Dates: First submitted 2011-05-24; First posted 2011-05-25 (Estimated); Last update posted 2012-11-14 (Estimated); Status verified 2012-11

CONDITIONS: Nonfatal Myocardial Infarction; Coronary Death
Keywords: MI; low dose aspirin; PPI; epidemiology; Nonfatal MI and coronary death

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Cases: Cases with nonfatal MI or coronary death
- Controls: Age, sex, and calendar-year matched controls sampled from the original study cohort to be a round number of at least four times the number of cases

SUMMARY:
The purpose of this study is to estimate the risk of myocardial infarction (MI)/coronary death associated with use of monotherapy low dose ASA (single antiplatelet) as well as concomitant use of monotherapy low dose ASA and proton pump inhibitors (PPIs) in patients with serious coronary heart disease using two UK primary care databases.

DETAILED DESCRIPTION:
Number of Anticipated Subjects: In case-control analysis: 10.000-15.000 participants

ELIGIBILITY:
Inclusion Criteria:

* As above ( study population description).
* All individuals aged 50-84 years with at least one year of enrolment with the primary care physician (PCP) and a computerized prescription history of at least one year before the start of the study.

Exclusion Criteria:

* Recorded diagnosis of cancer prior to study start.
* Patients aged ≥ 70 years with a follow-up longer than one year if having fewer than two recorded consultations with a primary care physician (PCP) during their entire follow-up (proxy for incomplete and invalid data recording

Ages: 50 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals aged 50-84 years who from 1 January 2000 to 31 December 2007 had a documented evidence of a hospitalization for a serious acute coronary event (MI, revascularization of coronary arteries or unstable angina) and who were alive 1 month after this event in two primary care clinical practice databases in the UK: General Practice Research Database (GPRD) and The Health Improvement Network (THIN).
Sampling Method: Non-Probability Sample
Enrollment: 42542 (Actual)
Dates: Start 2011-07; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Nonfatal MI or coronary death | Up to eight years from entry into study cohort

CONTACTS AND LOCATIONS:
Overall Officials: Luis A Garcia Rodriguez, Principal Investigator — CEIFE (Centro Español de Investigación Farmacoepidemiológica)
Locations (2):
- Research Site, Madrid, Spain
- Research Site, Mölndal, Sweden